CLINICAL TRIAL: NCT04582916
Title: PET Imaging of Cyclooxygenase in Participants With Major Depressive Disorder (MDD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 200157; 20-M-0157
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01-26

CONDITIONS: Depression
Keywords: PET Imaging; Inflammation; Cyclooxygenase-2; Depression
MeSH Terms: conditions — Depression; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- One Arm (Other): All subject receive the same tests
  Interventions: Drug: 11C-MCI; Drug: 11CPS13

INTERVENTIONS:
Drug: 11C-MCI — Injected IV followed by PET scanning
Drug: 11CPS13 — Injected IV followed by PET scanning

SUMMARY:
Background:

Researchers developed [11C]MC1, a radioligand for cyclooxygenase-2 (COX-2). COX-2 is an enzyme induced in the brain during inflammation. Researchers want to see the levels of COX-1 (measured as distribution volume VT) are elevated in the brain of two groups of mood disorders patients undergoing MDE relative to the control group.

Objective:

To determine whether COX-1 and COX-2 are detectable in the brains of individuals with MDD experiencing a major depressive episode (MDE).

Eligibility:

People aged 18-70 years with MDD and Healthy Volunteers aged 18 70 years.

Design:

Group A: MDD participants will be studied with the same dose of [11C]MC1 before and after administration of 600 mg celecoxib; the study is neither randomized nor placebo-controlled. Group B: MDD participants, both medicated and unmedicated, will be studied with [11C]PS13 and compared to healthy volunteers..

https://nimhcontent.nimh.nih.gov/start/surveys/?s=TJW4RA4WN3LDD988

DETAILED DESCRIPTION:
Study Description: This study will examine whether cyclooxygenase 1 (COX-1) and cyclooxygenase-2 (COX-2) are detectable in the brain of individuals with major depressive disorder (MDD).

Objectives: Primary Objective: To determine whether COX-1 and COX-2 are detectable in the brains of individuals with MDD experiencing a major depressive episode (MDE).

Endpoints: Primary Endpoints: Group A - Calculation of COX-2 density from [11C]MC1 PET scans, using baseline scans and scans after blockade with celecoxib. Group B - Calculation of the density of COX-1 using [11C]PS13

Secondary Endpoints, common to both groups:

1. the relationship between peripheral markers of inflammation and COX binding;
2. the relationship between clinical rating scales and COX binding

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients: In order to be eligible for this study, MDD participants must meet all of the following criteria:

1. Aged 18 to 70 years old.
2. Female participants of childbearing potential must be using a medically acceptable means of contraception.
3. Participants must be in good general health as evidenced by medical history and physical examination.
4. Each participant must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
5. All participants must have undergone a screening assessment under protocol 01M0254, The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Participants .
6. Participants must fulfill DSM-5 criteria for major depression (MDD) without psychotic features, as based on clinical assessment and structured diagnostic interview (SCID-P).
7. Participants must have an initial score on the MADRS greater than or equal to 18 or HAM-D greater than or equal to 15 within one week of study entry.
8. Participants must be experiencing an MDE lasting at least four weeks.
9. Unmedicated participants in both Groups must be medication-free for at least two weeks (5 weeks for aripirazole, brexpiprazole, fluoxetine) prior to first screen visit. Medications will not be discontinued for the purpose of this study.
10. Participants must have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
11. Participants must agree to adhere to the lifestyle considerations.

Healthy Controls: In order to be eligible to participate in this study, control subjects must meet all of the following criteria:

1. Aged 18 to 70 years old.
2. Female participants of childbearing potential must be using a medically acceptable means of contraception.
3. Able to provide informed consent.
4. Be in good general health, as evidenced by medical history and physical examination, and have no cognitive impairment.
5. Be enrolled in 01M0254, The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers or 17M0181, Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies .
6. Have their radial artery pulse checked for the presence of adequate ulnar collateral flow and the absence of any metal or foreign objects in both wrists.
7. Agree to adhere to the lifestyle considerations.

EXCLUSION CRITERIA:

Participants with MDD who meet any of the following criteria will be excluded from participation in this study:

1. Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen). Any lab value that is two-times the upper limit or even lower values in the investigator s judgment. Creatinine level >1.3 mg/dL.
2. Participants must be free of all prohibited medications or at least two weeks (5 weeks for aripiprazole, brexpiprazole, fluoxetine) prior to screen visit. These medications include antidepressants, anti-inflammatory drugs (except for study medication celecoxib), antipsychotics, anxiolytics, psychotropic drugs not otherwise specified (including herbal products), and sedatives/hypnotics. Medicated participants in Group B may continue their therapy.
3. Participants should not have taken Non-Steroidal Anti-Inflammatory Drug (NSAID)s for two weeks prior to the PET scan. Aspirin, corticosteroids (with the exception of topical steroids), or immunosuppressants (e.g. methotrexate) must not have been taken in the prior month.
4. Current psychotic features or a diagnosis of schizophrenia or any other psychotic disorder as defined in the DSM-5.
5. Participants with a history of DSM-5 substance use disorder (except for caffeinei or nicotine dependence) within the preceding three months. In addition, participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function of daily lfe.
6. Participants who, in the investigator s judgment, pose a current serious suicidal or homicidal risk.
7. Participants who have a history of aggressive behavior towards others.
8. Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
9. Participants seeking treatment or a change in treatment and may be referred to the community or to another research study.
10. Are unable to travel to the NIH.
11. Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
12. Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
13. Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
14. Pregnancy.
15. HIV Infection.
16. Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

Healthy controls who meet any of the following criteria will be excluded from participation in this study:

1. Clinically significant abnormalities on EKG or laboratory testing. This includes CBC and acute care panel (Na, K, Cl, CO2, creatinine, glucose, urea nitrogen).
2. Participants must be free of all prohibited medications or at least two weeks (5 weeks for aripiprazole, brexpiprazole, fluoxetine) prior to screen visit. These medications include antidepressants, anti-inflammatory drugs (except for study medication celecoxib), antipsychotics, anxiolytics, psychotropic drugs not otherwise specified (including herbal products), and sedatives/hypnotics.
3. Participants should not have taken NSAIDs for two weeks prior to the PET scan. Aspirin, corticosteroids, or immunosuppressants (e.g. methotrexate) must not have been taken in the prior month.
4. Participants with a history of DSM-5 substance use disorder (except for caffeine or nicotine dependence) within the preceding three months. In addition, participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function of daily life.
5. Participants who have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., an active infection or untreated malignancy).
6. Are unable to travel to the NIH.
7. Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits.
8. Have an inability to lie flat and/or lie still on the camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with the participant during the screening visit.
9. Are unable to have an MRI scan (e.g., because of pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, shrapnel fragments, or metal fragments in the eye.
10. Pregnancy.
11. HIV Infection.
12. Be NIMH staff or an NIH employee who is a subordinate/relative/co-worker of the investigators.

EXCLUSION OF CHILDREN:

Because this protocol has more than minimal risk from radiation exposure without possibility of direct benefit, inclusion of children is not appropriate.

EXCLUSION OF PREGNANT OR BREASTFEEDING WOMEN:

Pregnant women will be excluded because this protocol involves exposure to ionizing radiation. Lactating women will be excluded because radioisotopes may be excreted in milk.

EXCLUSION OF PARTICIPANTS WHO ARE HIV POSITIVE:

Persons with HIV infection are excluded because HIV infection itself may cause neuroinflammation, and we wish to specifically study the effect of depression on neuroinflammation.

EXCLUSION OF NON ENGLISH SPEAKING PARTICIPANTS:

Non-English-speaking participants will be excluded from participation in this study because neuropsychological testing is required by this protocol. This testing, which is critical for interpreting study results, has not been validated in other languages or when using a translator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2029-10-03 (Estimated); Study Completion 2030-04-11 (Estimated)

PRIMARY OUTCOMES:
Measure the concentration of radioligands | 36 months
  Tracer binding level

SECONDARY OUTCOMES:
measure peripheral markers of inflammation and COX binding | 36 months
  Assess the severity of depression and/or anxiety
measure clinical rating scales and COX binding | 36 months
  Assess the severity of depression and/or anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-M-0157.html